CLINICAL TRIAL: NCT00211549
Title: A Double-Blind, Placebo-Controlled Evaluation of the Safety and Efficacy of Three Doses of IDEA-033 in Comparison to Oral Naproxen for the Treatment of the Signs and Symptoms of Osteoarthritis of the Knee
Brief Title: An Effectiveness and Safety Study of IDEA-033 in Comparison to Oral Naproxen and Placebo for the Treatment of Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IDEA AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-033-III-04; NCT00371917 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

INTERVENTIONS:
Drug: IDEA-033

SUMMARY:
The purpose of this study is to identify the dose(s) of IDEA-033 that will provide a meaningful effect for treating osteoarthritis of the knee.

DETAILED DESCRIPTION:
The objective of this double-blind, placebo-controlled, randomized study is to evaluate the safety of and to identify the dose(s) of IDEA-033 that will provide a minimum clinically meaningful effect for treating the signs and symptoms of osteoarthritis of the knee. This study will also compare the safety profile of the three doses of IDEA-033 in treating the signs and symptoms associated with osteoarthritis for 12 weeks. The primary hypothesis is that at least one of the three doses of IDEA-033 is superior to placebo with respect to three primary efficacy endpoints of WOMAC Pain, WOMAC Physical Function, and Subject Global Assessment of Response to Therapy. A second hypothesis is that there is an increase in efficacy with increasing doses of IDEA-033.

Patients will receive one of five treatments for 12 weeks:Three doses of IDEA-033, or naproxen 1 g over-encapsulated tablet + placebo or placebo

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of both knees for minimum of six months
* Moderate pain in the most involved knee when not taking NSAIDs
* Must have used an oral NSAID on at least three days per week for last three months or 25 of 30 days before screening
* Demonstrate x-ray evidence of osteoarthritis in the most involved knee during the last six months

Exclusion Criteria:

* Grade 1 or Grade 4 severity of the most involved knee based on x-ray criteria
* Intra-articular injections or arthroscopy of the most involved knee during three months before Screening visit
* Inflammation of the most involved knee that could be related to gout or pseudogout-induced synovitis or infection
* A large bulging effusion
* History of gout or pseudo-gout induced synovitis or infection of the more severe knee
* History of partial or total knee replacement in either knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 875
Dates: Start 2005-06

PRIMARY OUTCOMES:
Change from baseline at Week 12 on pain subscale and physical function subscale on the WOMAC Osteoarthritis Index. Subject global assessment of response to therapy (SGART) on a five-point Likert scale at Week 12.

SECONDARY OUTCOMES:
Change from baseline at Weeks 2, 6, 9 for WOMAC pain and physical function scores and SGART. Mean change from baseline for the entire on-therapy period for WOMAC pain and physical function scores and SGART.

CONTACTS AND LOCATIONS:
Overall Officials: IDEA AG Clinical Trial, Study Director — IDEA AG
Locations (91):
- United States (91):
  - Birmingham, Alabama
  - Montgomery, Alabama
  - Drug Research and Analysis Corporation, Montgomery, Alabama
  - Northport, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Anaheim, California
  - Encinitas, California
  - Fair Oaks, California
  - Garden Grove, California
  - Irvine, California
  - Paramount, California
  - Rancho Mirage, California
  - San Diego, California
  - Spring Valley, California
  - Temecula, California
  - Vista, California
  - Northglenn, Colorado
  - Danbury, Connecticut
  - Clearwater, Florida
  - Coral Gables, Florida
  - Daytona Beach, Florida
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Ocala, Florida
  - Ocoee, Florida
  - Palm Harbor, Florida
  - Pembroke Pines, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Evansville, Indiana
  - Arkansas City, Kansas
  - Kansas City, Kansas
  - Newton, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Towson, Maryland
  - Milford, Massachusetts
  - East Lansing, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Flowood, Mississippi
  - Jackson, Mississippi
  - Kansas City, Missouri
  - Bozeman, Montana
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Dover, New Jersey
  - Binghamton, New York
  - Manilus, New York
  - Rochester, New York
  - Durham, North Carolina
  - Cumberland Research Associates L L C, Fayetteville, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Community Research Managment Associates, Cincinnati, Ohio
  - Colombus, Ohio
  - Columbus, Ohio
  - Franklin, Ohio
  - Perrysburg, Ohio
  - Bethany, Oklahoma
  - Beaver, Pennsylvania
  - Bensalem, Pennsylvania
  - Duncansville, Pennsylvania
  - Harleysville, Pennsylvania
  - Levittown, Pennsylvania
  - Penndel, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greer, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Spokane, Washington
  - Glendale, Wisconsin